CLINICAL TRIAL: NCT02356913
Title: A Pilot, Open Label, Randomised, Single Dose, Four-Period, Four-Treatment, Four-Sequence, Four Way Crossover Comparative Pharmacokinetic Study of Three Different 4 mg Nicotine Chewing Gum Test Formulations of Fertin Pharma A/S, Denmark With Nicorette Freshmint 4 mg Medicated Chewing Gum of McNeil Denmark ApS as Reference Formulation in Healthy, Adult, Human Smokers Under Fasting Conditions
Brief Title: Comparison of Pharmacokinetic Profiles of 3 New Nicotine Gum Formulations With a Reference Gum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fertin Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F-IN112; NIC/2013/1012 (Other: Fertin Pharma protocol ID number)
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Chewing Gum

ARMS (4):
- Gum A (Experimental): 4 mg nicotine gum; single dose; chewed 30 minutes
  Interventions: Drug: Nicotine gum
- Gum B (Experimental): 4 mg nicotine gum; single dose; chewed 30 minutes
  Interventions: Drug: Nicotine gum
- Gum C (Experimental): 4 mg nicotine gum; single dose; chewed 30 minutes
  Interventions: Drug: Nicotine gum
- Nicorette Freshmint (Active Comparator): 4 mg nicotine gum; single dose; chewed 30 minutes
  Interventions: Drug: Nicotine gum

INTERVENTIONS:
Drug: Nicotine gum

SUMMARY:
The purpose of the study is to compare the pharmacokinetic (PK) profiles and assess bioequivalence between three new nicotine gum formulations and a reference nicotine gum in healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, human smoker volunteers of any race within the age between 18 to 55 years.
* Willingness to provide informed consent to participate in the study
* Body Mass Index (BMI)> 18.5 kg/m2 to < 28.0 kg/m2.
* Smoke 5-10 cigarettes per day continuously for the last three (3) months
* Exhaled carbon monoxide ≥ 10 ppm at screening visit
* Successfully complete the training session
* Medically healthy subjects with clinically normal laboratory profiles, vital signs and ECGs as deemed by the Clinical Investigator
* Subject who are not in the process of quitting smoking
* Hemoglobin: ≥12.0 gm% for male and ≥11.5 gm% for female
* Absence of disease markers of HIV I & II, HBsAg, HCVAb and P24 antigen test.
* Females of childbearing age must be practicing an acceptable form of birth control for at least six months before screening and continue practicing an acceptable form of birth control during the study, unless they have had bilateral oophorectomy or tubal ligation or male partner has had vasectomy.
* Females of childbearing age agree to use acceptable form of birth control until the drug is washed out from the body i.e. 3 days after last dosing, unless male partner has had vasectomy.
* Absence of significant disease or clinically significant abnormal laboratory values on the laboratory evaluations, medical history or physical examination during the screening.
* Have a normal 12-lead ECG or one with abnormality considered clinically insignificant.
* Have a normal chest X-ray (P. A. view).
* Comprehension of the nature and purpose of the study and willingness to comply with the requirements of the entire procedure.
* Negative Breath alcohol test at every check in.
* Negative serum β-HCG at the time of screening and at every check in (for females only).
* Negative urine drug of abuse test (Barbiturates, Benzodiazepines, Opioids, Cocaine, Cannabinoids and Amphetamine, etc.) at every check-in. (This test will be done at the clinical facility).
* Willing to use Nicotine chewing gum during the study

Exclusion Criteria:

* History or presence of; drug abuse within the past year; hypersensitivity or idiosyncratic reaction to Nicotine or the resin of the gum preparation; any form of oral and/or pharyngeal inflammation; any form of oral lesions and/or gum disease or temperomandibular joint dysfunction; dentures or any dental work that could, in the opinion of the Investigator, affect the conduct of the study (including missing molars);
* Any major illness in the last three months or any significant ongoing chronic medical illness.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* Active deep vein thrombosis, arterial thromboembolic disorders or a history of these conditions
* History of or current gastro-intestinal diseases influencing drug absorption.
* Subjects who had been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Those who have used tobacco or nicotine containing products within 24 hours prior to the study drug administration on each study day.
* Subjects with carbon monoxide levels greater than or equal to 8 ppm in the morning prior to dosing.
* Suffer from xerostomia (dry mouth).
* Subjects using any smoking cessation aids such as nicotine replacement therapy (NRT), buproprion or varenicline during the last 3 months.
* History of neuropsychiatric diseases.
* History of breast cancer, endometrial cancer or other estrogen-dependent neoplasia, endometriosis and undiagnosed vaginal bleeding (for females only).
* Consumption of xanthine containing food and beverages [chocolates, tea, coffee or cola drinks] less than 48.0 hours prior to check in.
* Consumption of grapefruit/ Seville orange, grapefruit/ Seville orange juice products and poppy- containing food and beverages less than 48.0 hours prior to every check in.
* History of alcoholism (more than two years), moderate drinkers (more than three drinks per day) or having consumed alcohol less than 48.0 hours prior to check in.
* Participation in any clinical trial within last three months.
* History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm.
* Donation of blood (one unit or 350 mL or more) within last three months prior to receiving the first dose of investigational products.
* Use of any prescription drug therapy or over the counter (OTC) drugs or herbal products within two weeks prior to receiving the first dose of study medication and during the study [includes catecolamines, theophylline, clozapine and ropinirol].
* Pregnant women
* Breast feeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The maximum observed nicotine concentration in plasma (Cmax) | 12 hours
The area under the plasma concentration vs. time curve until the last measurable concentration (AUC0-t) | 12 hours
The area under the plasma concentration vs. time curve until infinity (AUC∞) | 12 hours

SECONDARY OUTCOMES:
Tmax | 12 hours from start of product administration
  The time of occurrence of Cmax following product administration
Kel | 12 hours
  The apparent Terminal Elimination Rate Constant of nicotine
T½ | 12 hours
  The apparent Terminal Elimination Half-life of nicotine
The amount of nicotine released from the gum during 30 minutes of chewing | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Tejas Acharya, M.D., Principal Investigator — Synchron Research Services Pvt. Ltd.